CLINICAL TRIAL: NCT01652469
Title: A Randomized Phase III Trial of Erlotinib Versus Docetaxel in Patients With Advanced Squamous Cell Non-small Cell Lung Cancer Who Failed First Line Platinum Based Doublet Chemotherapy Stratified by VeriStrat Good vs VeriStrat Poor
Brief Title: Testing of Drugs Erlotinib and Docetaxel in Lung Cancer Patients Classified Regarding Their Outlook Using VeriStrat®.
Acronym: EMPHASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP3-12; 2012-001896-35 (EudraCT Number)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: squamous cell; NSCLC; TKI; Erlotinib; Docetaxel; VeriStrat; protein signature
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Erlotinib (Experimental): Erlotinib in standard dose. Until progression (clinical or radiological) or unacceptable toxicity.
  Interventions: Drug: Erlotinib
- B: Docetaxel (Experimental): Docetaxel in standard dose. Until progression (clinical or radiological) or unacceptable toxicity.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg/day p.o. continuously with 21 days cycle.
  Other Names: Tarceva (Roche)
  Arms: A: Erlotinib
Drug: Docetaxel — Docetaxel 75 mg/m2 as an IV infusion every 21 days.
  Other Names: Taxotere (Sanofi-Aventis)
  Arms: B: Docetaxel

SUMMARY:
Using a laboratory test (VeriStrat), patients with relapsed squamous cell lung cancer are assigned to two strata, VSG (VeriStrat Good) and VSP (VeriStrat Poor). They are then randomized between an EGFR-TK inhibitor (erlotinib) and chemotherapy (Docetaxel).

It is hypothesized that the VeriStrat test results are able to predict the benefit of treatment with erlotinib vs docetaxel. This would suggest a significant improvement in progression-free survival for VSG patients when treated with Erlotinib, and no significant improvement in VSP patients who receive the same treatment.

DETAILED DESCRIPTION:
Goals of the study:

1. Explore the predictive ability of the VeriStrat signature, by testing for interaction between treatment arms (Arm A: erlotinib vs Arm B: docetaxel) and VeriStrat status (VSG vs VSP) using as outcome progression free survival.
2. Explore whether treatment with erlotinib provides progression free survival benefit as compared to docetaxel in the VSG group.
3. Compare progression free survival in the two treatment arms (Arm A: erlotinib vs Arm B: docetaxel) in the VSP group.
4. Explore the prognostic ability of the VeriStrat signature by testing for an overall difference in progression free survival between the two VeriStrat groups (in case of no significant interaction).
5. Explore the predictive ability of the VeriStrat signature using the secondary measures of clinical efficacy including overall survival, objective response rate, and disease control rate.
6. Compare overall survival, objective response rate and disease control rate between treatment groups separately in the VSG and VSP groups.
7. Explore the prognostic ability of the VeriStrat signature by testing for an overall difference in overall survival, objective response rate and disease control rate between the two VeriStrat groups (in case of no significant interaction).
8. Assess the safety and the tolerability of the two treatments separately in each VeriStrat group and overall.

Recruitment period: 18 months Sample Size: 500

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced stage IIIB, not amenable to radical radiotherapy, or metastatic stage IV non-small cell lung cancer (NSCLC) of predominant squamous subtype, according to the 7th edition of the TNM classification, including M1a (separate tumor nodule in a contralateral lobe, tumor with pleural nodules or malignant pleural or pericardial effusion) and/or M1b (distant metastasis).
* Progressive disease upon or after previous chemotherapy including at least one line of platinum-based chemotherapy.
* Measurable or evaluable disease according to RECIST v1.1 (Appendix 2).
* ECOG PS 0-2.
* Age ≥ 18 years.
* Adequate organ function, including:
* Adequate bone marrow reserve: ANC > 1.5 x 109/L, platelets > 100 x 109/L.
* Hepatic: bilirubin <1.5 x ULN; AP, ALT < 3.0 x ULN; AP, ALT <5 x ULN is acceptable in case of liver metastasis.
* Renal: calculated creatinine clearance > 40 ml/min based on the Cockroft and Gault formula.
* Signed and dated informed consent form.
* Male and female patients with reproductive potential must use an approved contraceptive method, during the trial and 12 months thereafter. Female patients with reproductive potential must have a negative pregnancy test within 7 days prior to study registration.
* Estimated life expectancy >12 weeks.
* Patient compliance and geographical proximity that allow adequate follow-up.

Exclusion Criteria:

* Evidence of other medical condition which would impair the ability of the patient to participate in the trial or might preclude therapy with trial drugs (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease, active infection, uncontrolled diabetes mellitus).
* Previous treatment with any EGFR-TKI or docetaxel.
* Documented brain metastases unless the patient has completed local therapy for central nervous system metastases and has been off corticosteroids for at least 14 days prior to study registration.
* Documented presence of activating EGFR mutations, if the patient was tested for EGFR mutations.
* Previous malignancy within the past 5 years with the exception of adequately treated cervical carcinoma in situ, breast cancer in situ or localized non-melanoma skin cancer.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with compliance for oral drug intake.
* Concurrent treatment with experimental drugs or other anti-cancer therapy treatment in a clinical trial within 21 days prior to study registration.
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs or any concomitant drugs contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD-PhD, Study Chair — Centre Pluridisciplinaire d'Oncologie, Centre Hospitalier Universitaire Vaudois, 1011 Lausanne, Switzerland; Egbert Smit, MD-PhD, Study Chair — Vrije Universiteit VU, Medical Centre, 1007MB Amsterdam, The Netherlands; Rolf Stahel, MD, Study Chair — Laboratory of Molecular Oncology, Clinic of Oncology, University Hospital Zürich, 8044 Zürich, Switzerland
Locations (32):
- Krankenhaus Hietzing, Vienna, Austria
- Institut Jules Bordet, Brussels, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- University Hospital of Heraklion, Heraklion, Greece
- National Institute of Oncology, Budapest, Hungary
- St James's Hospital, Dublin, Ireland
- Israel (2):
  - Institution Rabin MC, Petah Tikwa
  - Tel-Aviv Medical Center, Tel Aviv
- Italy (2):
  - Medical Oncology, Second University Naples, Naples
  - Vercelli Teaching Hospital, Vercelli
- Free University Medical Center, Amsterdam, Netherlands
- Spain (13):
  - Hospital general de Alicante, Alicante
  - Hospital Clínic Barcelona, Barcelona
  - Institut Català d'Oncologia - L'Hospitalet, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Ciudad Real General University Hospital, Ciudad Real
  - Onkologikoa, Donostia / San Sebastian
  - Hospital Severo Ochoa, Leganés
  - Hospital 12 de Octubre, Madrid
  - Carlos Haya Hospital, Málaga
  - Hospital Universitari Sant Joan, Reus
  - Hospital Arnau Vilanova Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
- Switzerland (6):
  - University Hospital Basel, Basel
  - Kantonsspital Graubünden, Chur
  - Fondation du centre Pluridisciplinaire d'Oncologie (CePO), Lausanne
  - Kantonsspital Luzern, Lucerne
  - Onkologiezentrum Berner Oberland, Thun
  - Universitätsspital Zürich, Zurich
- United Kingdom (2):
  - University Hospital South Manchester, Manchester
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Maio M, Chiodini P, Georgoulias V, Hatzidaki D, Takeda K, Wachters FM, Gebbia V, Smit EF, Morabito A, Gallo C, Perrone F, Gridelli C. Meta-analysis of single-agent chemotherapy compared with combination chemotherapy as second-line treatment of advanced non-small-cell lung cancer. J Clin Oncol. 2009 Apr 10;27(11):1836-43. doi: 10.1200/JCO.2008.17.5844. Epub 2009 Mar 9. PMID 19273711
- [Background] Shepherd FA, Dancey J, Ramlau R, Mattson K, Gralla R, O'Rourke M, Levitan N, Gressot L, Vincent M, Burkes R, Coughlin S, Kim Y, Berille J. Prospective randomized trial of docetaxel versus best supportive care in patients with non-small-cell lung cancer previously treated with platinum-based chemotherapy. J Clin Oncol. 2000 May;18(10):2095-103. doi: 10.1200/JCO.2000.18.10.2095. PMID 10811675
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Taguchi F, Solomon B, Gregorc V, Roder H, Gray R, Kasahara K, Nishio M, Brahmer J, Spreafico A, Ludovini V, Massion PP, Dziadziuszko R, Schiller J, Grigorieva J, Tsypin M, Hunsucker SW, Caprioli R, Duncan MW, Hirsch FR, Bunn PA Jr, Carbone DP. Mass spectrometry to classify non-small-cell lung cancer patients for clinical outcome after treatment with epidermal growth factor receptor tyrosine kinase inhibitors: a multicohort cross-institutional study. J Natl Cancer Inst. 2007 Jun 6;99(11):838-46. doi: 10.1093/jnci/djk195. PMID 17551144
- [Background] Yildiz PB, Shyr Y, Rahman JS, Wardwell NR, Zimmerman LJ, Shakhtour B, Gray WH, Chen S, Li M, Roder H, Liebler DC, Bigbee WL, Siegfried JM, Weissfeld JL, Gonzalez AL, Ninan M, Johnson DH, Carbone DP, Caprioli RM, Massion PP. Diagnostic accuracy of MALDI mass spectrometric analysis of unfractionated serum in lung cancer. J Thorac Oncol. 2007 Oct;2(10):893-901. doi: 10.1097/JTO.0b013e31814b8be7. PMID 17909350
- [Background] Sargent DJ, Conley BA, Allegra C, Collette L. Clinical trial designs for predictive marker validation in cancer treatment trials. J Clin Oncol. 2005 Mar 20;23(9):2020-7. doi: 10.1200/JCO.2005.01.112. PMID 15774793
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- See also: Related information — http://www.etop-eu.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Discrepancy between nb of enrolled pts and nb of pts who started treatment,because 1 patient,who shouldn't have been included (exclusion criteria),was enrolled in the database by mistake.In the database patient's status couldn't be changed from "Enrolled" to "Ineligible",thus this patient considered enrolled,but was not included in efficacy cohort.
Period: Overall Study
Arm/Group | A: Erlotinib | B: Docetaxel
Started | 38 | 42
Completed | 37 | 36
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Erlotinib | B: Docetaxel | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Median (Full Range); unit: years] | 66.7 [44.4 to 81.9] | 70.1 [53.3 to 84.0] | 68.7 [44.4 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 31 | 35 | 66
Smoking history [Count of Participants; unit: Participants]
  Current | 16 | 12 | 28
  Former (>100 cigarettes & >12 months smoke-free) | 20 | 28 | 48
  Never | 2 | 2 | 4
ECOG performance status [Count of Participants; unit: Participants] — ECOG Performance status scaling:
  PS 0:Fully active, able to carry on all pre-disease performance without restriction PS 1:Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work PS 2:Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours PS 3:Capable of only limited self-care, confined to bed or chair more than 50% of waking hours PS 4:Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  Participants
    0 | 12 | 15 | 27
    1 | 24 | 22 | 46
    2 | 2 | 5 | 7
VeriStrat status [Count of Participants; unit: Participants]
  Good | 28 | 30 | 58
  Poor | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from the date of randomization until documented progression or death without documented progression.
  Assessment of Progressive Disease (PD) based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) Target lesions:At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.(Note: the appearance of one or more new lesions is also considered progression).
  Non-target lesions:Unequivocal progression of existing non-target lesions. (Note:the appearance of one or more new lesions is also considered progression). To achieve 'unequivocal progression', there must be an overall level of substantial worsening in non-target disease such that,even in presence of SD or PR in target disease, the overall tumour burden has increased sufficiently
Time Frame: The combined run in period, treatment and follow-up for PFS is expected to extend the study duration to a total of 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Erlotinib | B: Docetaxel
Number analyzed (Participants) | 38 | 42
months | 1.6 [1.3 to 3.8] | 3.0 [1.9 to 4.2]

2. Secondary Outcome: Overall Survival
Description: Defined as time from the date of randomization until death from any cause.
Time Frame: All patients will be followed for survival status every 12 weeks up to 24 months after the last patient is randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A: Erlotinib | B: Docetaxel
Number analyzed (Participants) | 38 | 42
months | 7.1 [4.4 to 10.6] | 7.1 [5.3 to 8.6]

3. Secondary Outcome: Objective Response
Description: Objective response is defined as best overall response (CR or PR) across all assessment time-points according to RECIST Criteria 1.1 during the period from randomization to termination of trial treatment.
Time Frame: Same as primary outcome: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: Erlotinib | B: Docetaxel
Number analyzed (Participants) | 38 | 42
Participants
  Partial response | 4 | 6
  Stable Disease | 15 | 18
  Progressive Disease | 17 | 14
  Non-Evaluable | 2 | 4

4. Secondary Outcome: Disease Control
Description: Disease control is defined as achieving objective response or stable disease for at least 6 weeks.
Time Frame: Same as primary outcome: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | A: Erlotinib | B: Docetaxel
Number analyzed (Participants) | 38 | 42
Participants
  Disease Control | 19 | 24
  No Disease Control | 19 | 18

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events classified according to NCI CTCAE version 4
Time Frame: Same as primary outcome: 24 months
Population: One patient from the Docetaxel arm never started treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Erlotinib | B: Docetaxel
Number analyzed (Participants) | 38 | 41
Participants
  Experienced AE/SAE | 36 | 39
  No AE/SAE | 2 | 2
  Experienced SAE | 7 | 19

ADVERSE EVENTS:
Description: One patient from the Docetaxel arm never started treatment.
Arm/Group | A: Erlotinib | B: Docetaxel
All-Cause Mortality (participants affected / at risk) | 7/38 | 3/41
Serious Adverse Events (participants affected / at risk) | 7/38 | 19/41
Other Adverse Events (participants affected / at risk) | 36/38 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Erlotinib (N=38) | B: Docetaxel (N=41)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6
Lung infection (Infections and infestations) | 2 | 2
Bronchial infection (Infections and infestations) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infections and infestations (Infections and infestations) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Erlotinib (N=38) | B: Docetaxel (N=41)
Fatigue (General disorders) | 11 | 24
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Diarrhea (Gastrointestinal disorders) | 10 | 11
Anorexia (Metabolism and nutrition disorders) | 7 | 8
Neutrophil count decreased (Investigations) | 2 | 12
Mucositis oral (Gastrointestinal disorders) | 5 | 9
Nausea (Gastrointestinal disorders) | 4 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 11
Pain (General disorders) | 4 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 1
Lung infection (Infections and infestations) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 4
Fever (General disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3
Edema limbs (General disorders) | 1 | 4
Flu-like symptoms (General disorders) | 2 | 3
Hypertension (Vascular disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 2
Aspartate aminotransferase increase (Investigations) | 3 | 1
Conjuctivitis (Eye disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Death NOS (General disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Creatinine increase (Investigations) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorders (Gastrointestinal disorders) | 2 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 3
Oral dysesthesia (Gastrointestinal disorders) | 2 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol (2012-05-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT01652469/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2015-01-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT01652469/SAP_002.pdf
  • Statistical Analysis Plan: moc figures SAP (2015-01-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT01652469/SAP_003.pdf
  • Statistical Analysis Plan: moc tables SAP (2015-01-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT01652469/SAP_004.pdf
  • Informed Consent Form (2012-05-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT01652469/ICF_001.pdf